CLINICAL TRIAL: NCT04825275
Title: Neuro-pharmacological Properties of Repurposed Posaconazole in Glioblastoma: A Phase 0 Clinical Trial
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to slow accrual.
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alireza Mansouri, Assistant Professor, Department of Neurosurgery, Penn State Health Milton S Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015948; 1R03CA255992-01 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain; Glioblastoma Multiforme, Adult
Keywords: Glioblastoma; Glioblastoma Multiforme; GBM; Brain cancer; Posaconazole; Anti-fungal agents
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posaconazole (Experimental): Participants will be taking 300 mg of the study drug (three 100 mg tablets) by mouth twice a day the first day and then 300 mg once a day until the day of biopsy or surgery. On the day of biopsy or surgery, participants will take their medication the morning of their biopsy or surgery (before the operation). Participants will then take the last dose of the medication in the morning of the day after their biopsy or surgery. Participants will be given 12 days' worth of the study drug (pills) and verbally instructed how and when to take them.
  Interventions: Drug: Posaconazole Pill
- Control (No Intervention): Participants will not undergo any intervention.

INTERVENTIONS:
Drug: Posaconazole Pill — 300 mg (three 100 mg tablets) orally
  Other Names: Noxafil
  Arms: Posaconazole

SUMMARY:
This research is being done to find out if the study drug (posaconazole) can enter brain tumors at a high enough amount to stop the tumor cells from dividing. Posaconazole is a drug which doctors already use for fungal infections and is thought to be able to effect tumor cells. As treatments for this type of brain tumor are limited, it is hoped that the results of this study will help to determine if the study drug should be studied further as a possible treatment.

DETAILED DESCRIPTION:
Both ketoconazole and posaconazole are FDA-approved anti-fungal agents with a well-established side effect and safety profile. Ketoconazole and posaconazole have shown efficacy in reducing tumor cell proliferation in in-vitro studies. Furthermore, both have also shown efficacy, mediated at least in part through inhibition of HK2 activity, in animal models with dosing concentration and schedules that are documented as safe in humans. As a drug, posaconazole has a more predictable half-life than ketoconazole and has less off-target effects. Therefore, the proposed trial will focus on the role of posaconazole exclusively. As a first step, demonstration of adequate penetrance of study drug in brain and tumor tissue (pharmacokinetics) and biological effect (inhibition of glycolysis and subsequent tumor cell death) is necessary prior to large scale clinical studies. A total of 5 control participants will be included in this study as the investigator specifically wants to assess for pharmacodynamic differences too. The addition of a control group to this study rather to both the studies (ketoconazole study is a separate protocol) is because the investigator feels posaconazole may be a more promising drug for moving forward.

Plasma drug concentration measurements are an unreliable method to assess delivery of drugs across the blood-brain barrier. In contrast, intracerebral MDC monitoring allows for approximate measurements within extracellular fluid (ECF) sampling of the brain. MDC placement within the brain is not a novel technique and has been utilized routinely in the ICU setting to measure brain metabolism by sampling of ECF of traumatic brain injury patients [59-61].

MDC are now FDA-approved and are being placed routinely with intracranial pressure monitors. This method allows for continuous measurement of ECF within a tumor or normal tissue. The dialysis probe has a semipermeable membrane which is less than 1 mm in diameter into which two sections of microcatheter are fused. Previous studies have demonstrated the feasibility of keeping the catheters in place of critically injured patients for up to 2 weeks [62-64].

When placed at the time of surgical resection, the microcatheters are stereotactically implanted, placing the probe within the desired brain and/or tumor region. Externally, the catheter is connected to a syringe pump, which delivers a low flow rate (μl/min) of continuous perfusion fluid (Lactated Ringers or artificial CSF) and dialysate is collected in a microvial from the outlet tube. This sterile, single use catheter is minimally invasive and developed to achieve optimal diffusing characteristics similar to passive diffusion of a capillary blood vessel. Just as in the function of brain capillary vessel, water, inorganic ions and small organic molecules freely diffuse across the membrane of the probe, whereas proteins and protein bound compounds are impermeable. Additionally, lipophilic compounds are poorly recovered. Therefore, assessment of pharmacokinetics of drug using MDC provides valuable insight relevant to its anti-neoplastic properties.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Evidence of primary or recurrent HGG that in the opinion of the treating team would require surgical resection
* Karnofsky Performance Score (KPS) ≥ 60%
* ECOG ≤ 2
* Life expectancy greater than 12 weeks
* Adequate liver function defined as ALT, AST, ALP within 1.5x institutional upper limit of normal (for study drug arm only)
* Ability to swallow medication (for study drug arm only)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation (for study drug arm only)
* Ability to understand and willingness to sign a written informed consent document
* Be able to comply with treatment plan, study procedures and follow-up examinations

Exclusion Criteria:

* Patients may not be receiving any other investigational agents while on study
* Patients who have known allergy to posaconazole or other azoles (for study drug arm only)
* Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous azole class drugs for a parasitic infection (for study drug arm only)
* Patients with a history of acute or chronic hepatitis (for study drug arm only)
* Patients with liver enzymes (ALT, AST, ALP) >1.5x above normal range for the laboratory performing the test (for study drug arm only)
* Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting posaconazole therapy (for study drug arm only)
* Patients who are taking any anti-convulsant medication that interferes with the cytochrome P450 pathway (e.g. phenytoin, phenobarbital, carbamazepine, etc.) and who cannot be switched to alternative medications such as keppra (levetiracetam) (for study drug arm only)
* Uncontrolled intercurrent illness such as chronic hepatitis, acute hepatitis, or psychiatric illness/social situation that would limit compliance with study requirements (for study drug arm only)
* Patients with a history of Addison's disease or other forms of adrenal insufficiency (for study drug arm only)
* Patient with little or no stomach acid production (achlorhydria) (for study drug arm only)
* Pregnant and breast feeding women)
* Patients with a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product administration or may interfere with the interpretation of the results.
* Patients who are not available for follow-up assessments or unable to comply with study requirements.
* Patients who are currently taking medications that induce the metabolism of posaconazole, such as isoniazid, nevirapine, rifamycins (such as rifabutin, rifampin), or St. John's wort and cannot be safely discontinued off of them for the duration of the trial (for study drug arm only).
* Patients who are currently taking medications for which the metabolism may be affected by posaconazole, which include but are not limited to: benzodiazepines (such as alprazolam, midazolam, triazolam), domperidone, eletriptan, eplerenone, ergot drugs (such as ergotamine), nisoldipine, drugs used to treat erectile dysfunction-ED or pulmonary hypertension (such as sildenafil, tadalafil), some drugs used to treat seizures (such as carbamazepine, phenytoin), some statin drugs (such as atorvastatin, lovastatin, simvastatin) (for study drug arm only).
* Patients who are non-English speakers
* Patients who are not capable of understanding the consent form and would need a legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Mansouri, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhanja D, Neighbors J, Connor J, Zadeh G, Mansouri A. Neuropharmacological Study of Posaconazole for Glioblastoma: A Phase 0 Clinical Trial Protocol. Neurosurgery. 2022 Oct 1;91(4):658-665. doi: 10.1227/neu.0000000000002071. Epub 2022 Jul 25. PMID 35861778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven participants gave informed consent to participate in the clinical trial. One participant withdrew consent prior to beginning dosing posaconazole.
Pre-assignment Details: Participants were assigned to the Control Arm if their tumor resection surgery was scheduled more than 7-10 days after informed consent was obtained.
Period: Overall Study
Arm/Group | Posaconazole | Control
Started | 3 | 4
Completed | 2 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole | Control | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 4 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Neuro-pharmacokinetic Profile of Posaconazole Prior to Dosing [Mean (Standard Deviation); unit: ng/mL] — Although it was impossible to obtain CSF to test the neuro-pharmacokinetic profile prior to implantation of the microdialysis catheter during tumor resection surgery (at which point participants were already dosed with posaconazole), participants taking azole drugs outside of the study prior to surgery were not included. So, the baseline neuro-pharmacokinetic profile of posaconazole is not applicable. Population: Since CSF was not collected prior to tumor resection surgery (or posaconazole dosing), the baseline neuro-pharmacokinetic profile of posaconazole is not applicable.

OUTCOME MEASURES:

1. Primary Outcome: Posaconazole Concentration in Cerebrospinal Fluid Using Microdialysis Catheters
Description: Assessment of the concentration of drug in the dialysate fluid.
Time Frame: Collected over a 24-hour period after surgery (biopsy or resection)
Population: The fourth control participant's samples were unavailable for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 3
ng/mL | NA (NA) — Results were less than the limit of detection. | NA (NA) — Results were less than the limit of detection.

2. Secondary Outcome: Number of Participants Able to Tolerate Preoperative Steady-state Dosing of Posaconazole
Description: Measured through the Grade and Frequency of adverse events, based on the CTCAE v5.0 criteria
Time Frame: from Baseline to Visit 7 (14 days +/- 7 days post-op)
Population: Control participants did not take the study drug.
Measure: Number; unit: Participants Who Tolerated Dosing
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 0
Participants Who Tolerated Dosing | 2 |

3. Secondary Outcome: Posaconazole Effect on Hexokinase 2 Concentration Within Tumor Tissue
Description: Measured using a hexokinase-2 ELISA with a range of 1.56 ng/mL - 100 ng/mL on tumor tissue.
Time Frame: Within 24 hours after biopsy or tumor resection
Population: The fourth control participant's samples were unavailable for analysis.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 3
ng/mg | NA (NA) — Results were all less than the limit of detection. | NA (NA) — Results were all less than the limit of detection.

4. Secondary Outcome: Posaconazole Effect on Tumor Proliferation in Tumor Tissue
Description: Measured using Ki-67 proliferation index with of a range of 0% proliferation (no proliferation) to 100% (high proliferation). Ki-67 is a marker found in actively dividing cells. A higher Ki-67 value may signify a more aggressive tumor. Ki-67 is routinely measured during pathology analysis of tumor samples.
Time Frame: Within 24 hours after biopsy or tumor resection
Measure: Mean (Standard Deviation); unit: % cells actively dividing
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 4
% cells actively dividing | 25 (0.05) | 39 (0.134)

5. Secondary Outcome: Posaconazole Effect on Cell Death in Tumor Tissue
Description: Measured using a BCL-2 ELISA with a range of 0.156 ng/mL to 10 ng/mL.
Time Frame: Within 24 hours after biopsy or tumor resection
Population: The fourth control participant's samples were unavailable for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 3
ng/mL | 0.3078 (0.2418) | 0.5363 (0.2908)

6. Secondary Outcome: Posaconazole Effect on Angiogenesis in Tumor Tissue
Description: Measured using a CD31 ELISA with a range of 31.2 pg/mL to 2000 pg/mL.
Time Frame: Within 24 hours after biopsy or tumor resection
Population: The fourth control participant's samples were unavailable for analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 2 | 3
pg/mL | 2130 (1500) | 2240 (499.8)

7. Secondary Outcome: Correlation of Neuro-pharmacokinetic Profile of Posaconazole With Lactate Concentration
Description: The concentration vs. time profile of posaconazole will be correlated with the concentration vs. time profile of lactate in the cerebrospinal fluid.
Time Frame: Collected over a 24-hour period after surgery (biopsy or resection)
Population: The entirety of the cerebrospinal fluid collected from the microdialysis catheters was consumed during the posaconazole concentration analysis. Since the catheters yielded a low volume of sample, none was available to test lactate concentration, thus, correlation of posaconazole profile to lactate concentration could not be analyzed for any of the participants.
Measure: Mean (Standard Deviation); unit: Correlation Coefficient
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlation of Neuro-pharmacokinetic Profile of Posaconazole With Pyruvate Concentration
Description: The concentration vs. time profile of posaconazole will be correlated with the concentration vs. time profile of pyruvate in the cerebrospinal fluid.
Time Frame: Collected over a 24-hour period after surgery (biopsy or resection)
Population: The entirety of the cerebrospinal fluid collected from the microdialysis catheters was consumed during the posaconazole concentration analysis. Since the catheters yielded a low volume of sample, none was available to test pyruvate concentration, thus, correlation of posaconazole profile to pyruvate concentration could not be analyzed for any of the participants.
Measure: Mean (Standard Deviation); unit: Correlation Coefficient
Arm/Group | Posaconazole | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the Baseline visit through Visit 7 (14+/-7 days Post-Op).
Arm/Group | Posaconazole | Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=2) | Control (N=4)
Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Hypertensive Emergency
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=2) | Control (N=4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Low HCT (Investigations) | 0 (0) | 1 (1)
Low RBC (Investigations) | 0 (0) | 1 (1)
Increased RDW (Investigations) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Renal Disorder - BUN Increased (Investigations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Asymptomatic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation in data analysis is failure to meet the enrollment goal. Enrollment was difficult due to the rare nature of the disease and the 7-10 day dosing window. Some patients were eligible, but immediate surgical intervention was necessary, so they could not reach steady-state posaconazole.

Two planned outcome measures, correlation of neuro-pharmacokinetic profile with concentration of lactate and pyruvate, were not analyzed due to limited volume of cerebrospinal fluid from microdialysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04825275/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04825275/ICF_001.pdf